CLINICAL TRIAL: NCT02967055
Title: The Effect of Isotretinoin on the Etonogestrel Contraceptive Implant
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0614
Record Dates: First submitted 2016-11-14; First posted 2016-11-17 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This exploratory study will fill a knowledge gap regarding the pharmacokinetic effects of isotretinoin on the etonogestrel (ENG) contraceptive implant.

DETAILED DESCRIPTION:
The Investigators will enroll only women with an etonogestrel contraceptive implant in place who are initiating isotretinoin therapy through their dermatologist. The Investigators will monitor the subjects serum etonogestrel concentration during isotretinoin therapy but no medications will be provided through this study. No medical devices will be inserted as part of this study either.

ELIGIBILITY:
Inclusion Criteria:

* Have a secondary form of non-hormonal contraception or abstain during isotretinoin therapy and four weeks afterwards
* Have at least two negative pregnancy tests at least 19 days apart prior to initiating isotretinoin therapy
* Have normal baseline laboratory evaluation including liver function tests, basic metabolic panel, and complete blood count
* Willing to abstain from taking any Vitamin A supplement during the study period
* Have a Body Mass Index (BMI) >= 18.5

Exclusion Criteria:

* Currently breastfeeding
* Known contraindications to isotretinoin
* Currently taking any known cytochrome P-450 3A4 enzyme inducers or inhibitors

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive-aged women (18-45) who are under the care of a dermatologist for treatment of acne and planning to initiate therapy with isotretinoin. The women must have chosen an ENG contraceptive implant for their primary mechanism of birth control, placed at least four weeks prior to study enrollment, but in place no longer than three years.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lazorwitz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled Participants: Participants meeting all inclusion/exclusion criteria and enrolled into the study
Period: Overall Study
Arm/Group | Enrolled Participants
Started | 54 (Assessed for eligibility)
In-person Screening (Presented for In-person screening) | 14
Enrolled | 9 (Enrolled)
Completed 4 Week Follow-up Visit | 8
Completed | 5
Not Completed | 49
Not completed — Excluded | 40
Not completed — Screen fail | 3
Not completed — Lost to Follow-up | 2
Not completed — Stopped due to side effects | 3
Not completed — Stopped due to drug cost | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 21 [18 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
Body-mass index [Median (Full Range); unit: kg/m^2] | 27.4 [21.1 to 34.9]

OUTCOME MEASURES:

1. Primary Outcome: Serum Etonogestrel (ENG) Level
Description: ENG levels will be measured prior to initiation of isotretinoin therapy.
Time Frame: Baseline (enrollment)
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 8
pg/mL | 243.3 [166.14 to 294.5]

2. Primary Outcome: Serum Etonogestrel (ENG) Level
Description: ENG levels will be measured 4 weeks after of initiation of isotretinoin therapy.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 8
pg/mL | 234.0 [185.0 to 256.9]

3. Primary Outcome: Serum Etonogestrel (ENG) Level
Description: ENG levels will be measured 9 weeks after of initiation of isotretinoin therapy.
Time Frame: 9 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 5
pg/mL | 145.4 [138.6 to 235.4]

ADVERSE EVENTS:
Time Frame: 20 weeks from onset of isotretinoin therapy
Description: Collected primarily any pregnancies
Arm/Group | Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02967055/Prot_SAP_000.pdf